CLINICAL TRIAL: NCT02148146
Title: Clinical Trial of Omegaven™ Therapy for Parenteral Nutrition Associated Cholestasis
Brief Title: Use of Omega 3 Oil Emulsion for Parenteral Nutrition Associated Cholestasis
Status: No longer available | Type: Expanded Access
Sponsor: University of California, San Diego (Other)
Responsible Party: Sponsor
Other Study IDs: 105591
Record Dates: First submitted 2014-05-20; First posted 2014-05-28 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Cholestasis
Keywords: short bowel syndrome; intestinal failure; total parenteral nutrition associated cholestasis
MeSH Terms: conditions — Cholestasis; Short Bowel Syndrome; Intestinal Failure | interventions — fish oil triglycerides

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Omegaven — Fish oil emulsion given 1g/kg/day as infusion

SUMMARY:
This is a clinical study designed to evaluate the safety and benefit of a fish oil based fat emulsion in the treatment of liver disease associated with prolonged use of intravenous nutrition.

DETAILED DESCRIPTION:
Specific Aims of Study

1. To determine the safety profile of an intravenous omega-3 fat emulsion (Omegaven™)
2. To determine if established PN associated liver disease can be reversed or its progression halted by using a parenteral fat emulsion prepared from fish oil as measured by normalization of serum levels of hepatic enzymes and bilirubin.

ELIGIBILITY:
Inclusion Criteria:

1. Age < 18 years old
2. Patients will be PN dependent (unable to meet nutritional needs solely by enteral nutrition) and are expected to require PN for at least another 30 days, may be inpatient or outpatient
3. Patients considered eligible for study participation must have parenteral nutrition associated liver disease (PNALD) as defined as a direct bilirubin of 2 mg/dl or more. Other causes of liver disease should be excluded. A liver biopsy is not necessary for treatment
4. Direct bilirubin > 2.0 mg/dl
5. Signed patient informed consent
6. The patient must have utilized standard therapies to prevent the progression of his/her liver disease including surgical treatment, cyclic PN, avoiding overfeeding, reduction/removal of copper and manganese from PN, advancement of enteral feeding, or the use of ursodiol (i.e., Actigall®)

Exclusion Criteria:

1. Pregnancy
2. Other causes of chronic liver disease (Hepatitis C, Cystic fibrosis, biliary atresia, and alpha 1 anti-trypsin deficiency)
3. Enrollment in any other clinical trial involving an investigational agent (unless approved by the designated physicians on the multidisciplinary team)
4. The parent or guardian or child unwilling to provide consent or assent
5. Patients known to be allergic to fish or egg protein and patients with the following contraindications to Omegaven™ use:

   * Impaired lipid metabolism
   * Severe hemorrhagic disorders
   * Unstable diabetes mellitus
   * Collapse and shock
   * Stroke/embolism
   * Recent cardiac infarction
   * Undefined coma status

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Lazar, MPH, Principal Investigator — UC San Diego Medical Center
Locations (2):
- United States (2):
  - UC San Diego Medical Center, San Diego, California
  - Rady Children's Hospital of San Diego, San Diego, California